CLINICAL TRIAL: NCT03199183
Title: Registration Study of Takayasu's Arteritis in China
Acronym: TA-China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-ZX43
Record Dates: First submitted 2017-06-23; First posted 2017-06-26 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Takayasu Arteritis
Keywords: Takayasu Arteritis; registry
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — All participants will have samples with DNA taken for laboratory biomarker analysis or genetic sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Takayasu arteritis: All recruited Takayasu arteritis patients.
  Interventions: Radiation: PET-CT; Other: laboratory biomarker analysis; Genetic: genetic sequencing

INTERVENTIONS:
Radiation: PET-CT — PET-CT will be proceed on the basis of clinical status and aspiration of individual patient. The imaging results will be analysed by professional radiologists.
Other: laboratory biomarker analysis — Screening of potential biomarkers related to Takayasu arteritis and verification tests will be operated.
Genetic: genetic sequencing — Genetic sequencing results will be analysed to identify susceptible alleles or single nucleotide polymorphisms of Takayasu arteritis.

SUMMARY:
Takayasu arteritis(TA) is a chronic progressive vasculitis predominantly affecting the aorta and its major branches. The demographic, clinical and prognostic features of Takayasu arteritis in China remains in uncertainties. Investigators aim to setup a national registration study for Takayasu arteritis, to observe the prevalence, clinical manifestations, natural history, survival, progression, diagnostic and therapeutic methods of the disease in China.

DETAILED DESCRIPTION:
Objective: The study aims to investigate the demographic, clinical and prognostic features and to draw the diagnostic and therapeutic algorithm of Takayasu arteritis in China.

Study Type: A national, multicenter, observational, ambispective cohort study.

Study Design: The cardinal contents of this registry study are as follows:

1. Select representative clinical centers through typical sampling methods and train the local investigators in basic knowledge of Takayasu arteritis. Introduce the Electronic Data Capture System and train in completing case report forms.
2. Collect demographic, clinical, imaging, laboratory, diagnostic and therapeutic information of Takayasu arteritis patients hospitalized from Jan 1st 2002 to now. Build a baseline database of Takayasu arteritis patients.
3. Recruit new diagnosed Takayasu arteritis patients in future 2 years from 2017 or till reaching a total of 1067 registered patients.
4. Gather the 3-month, 6-month, 1-year follow up information including general, clinical, therapeutic, prognostic data of all recruits and build up the follow-up database.
5. Establish bio-bank for serum/plasma, urine, stool, tissues or cells.

Data management, quality control and statistic analysis: Electronic Data Capture System has been built and the investigators will manage and analyze data in align with key indicators. The investigators have invited professional statistic analysts to assist analyzing data and a third party to supervise data quality.

Ethics: The Ethics Committee of Fuwai Hospital approved this study and following ethical supports from participating centers are required. Informed consents before patient enrollment are required.

ELIGIBILITY:
Inclusion Criteria:

All of the patients diagnosed in participating clinical centers with Takayasu arteritis fulfilled the American College of Rheumatology 1990 criteria for the classification of Takayasu arteritis or the 1996 revised diagnostic criteria for Takayasu arteritis from Ishikawa K by Sharma BK et al. Patients highly suspected as Takayasu arteritis but uncertain in local centers can apply for assistant diagnosis of senior medical institutions.

Exclusion Criteria:

1. Manifestations caused by other diseases: atherosclerosis, fibromuscular dysplasia, Bechet's disease, giant cell arteritis, congenital vascular malformation, syphilis and other infections resulting in vasculitis.
2. Pregnant women and lactating women.
3. None indications for Takayasu arteritis from ultrasound, computed tomographic angiography, magnetic resonance angiography, digital subtraction angiography.
4. Absence of patient consents or dropout during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Takayasu arteritis patients diagnosed in all participant centers.
Sampling Method: Non-Probability Sample
Enrollment: 1067 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
prevalence rate | 1 year
  the percentage of Takayasu arteritis patients among general population (estimated) during one-year period

SECONDARY OUTCOMES:
survival rate or mortality rate | 1 year, at 3-month interval
  the percentage of alive or dead recruits
rehospitalization rate | 1 year, at 3-month interval
  the percentage of readmission to hospitals or centers

CONTACTS AND LOCATIONS:
Overall Officials: Huimin Zhang, MD., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Jun Cai, MD.PhD., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Consent for sharing of non identifiable study data for regulatory authorities.

REFERENCES:
- [Background] Ishikawa K. Diagnostic approach and proposed criteria for the clinical diagnosis of Takayasu's arteriopathy. J Am Coll Cardiol. 1988 Oct;12(4):964-72. doi: 10.1016/0735-1097(88)90462-7. PMID 2901440
- [Background] Arend WP, Michel BA, Bloch DA, Hunder GG, Calabrese LH, Edworthy SM, Fauci AS, Leavitt RY, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Takayasu arteritis. Arthritis Rheum. 1990 Aug;33(8):1129-34. doi: 10.1002/art.1780330811. PMID 1975175
- [Background] Yang L, Zhang H, Jiang X, Zou Y, Qin F, Song L, Guan T, Wu H, Xu L, Liu Y, Zhou X, Bian J, Hui R, Zheng D. Clinical manifestations and longterm outcome for patients with Takayasu arteritis in China. J Rheumatol. 2014 Dec;41(12):2439-46. doi: 10.3899/jrheum.140664. Epub 2014 Oct 1. PMID 25274886
- [Background] Sharma BK, Jain S, Suri S, Numano F. Diagnostic criteria for Takayasu arteritis. Int J Cardiol. 1996 Aug;54 Suppl:S141-7. doi: 10.1016/s0167-5273(96)88783-3. PMID 9119516
- [Derived] Fan L, Yang L, Wei D, Ma W, Lou Y, Song L, Bian J, Zhang H, Cai J. Clinical Scenario and Long-Term Outcome of Childhood Takayasu Arteritis Undergoing 121 Endovascular Interventions: A Large Cohort Over a Fifteen-Year Period. Arthritis Care Res (Hoboken). 2021 Nov;73(11):1678-1688. doi: 10.1002/acr.24387. Epub 2021 Oct 13. PMID 32702156
- [Derived] Fan L, Zhang H, Cai J, Yang L, Wei D, Yu J, Fan J, Song L, Ma W, Lou Y. Clinical Course, Management, and Outcomes of Pediatric Takayasu Arteritis Initially Presenting With Hypertension: A 16-year overview. Am J Hypertens. 2019 Sep 24;32(10):1021-1029. doi: 10.1093/ajh/hpz103. PMID 31278892
- [Derived] Fan L, Zhang H, Cai J, Yang L, Liu B, Wei D, Yu J, Fan J, Song L, Ma W, Zhou X, Wu H, Lou Y. Clinical course and prognostic factors of childhood Takayasu's arteritis: over 15-year comprehensive analysis of 101 patients. Arthritis Res Ther. 2019 Jan 22;21(1):31. doi: 10.1186/s13075-018-1790-x. PMID 30670069